CLINICAL TRIAL: NCT00351546
Title: A Study to Assess the Effects of DPP-4 Inhibition on Insulin Sensitivity in Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2352
Record Dates: First submitted 2006-07-11; First posted 2006-07-13 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Vildagliptin; Type 2 diabetes; Insulin sensitivity; Insulin action
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Vildagliptin

INTERVENTIONS:
Drug: Vildagliptin

SUMMARY:
Type 2 diabetes results when the body does not produce enough insulin and/or is unable to properly use the insulin it makes (insulin resistance). This study was undertaken to assess the effects of vildagliptin on insulin sensitivity in people with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes at least 3 months prior to screening
* Blood glucose criteria must be met
* On stable dose of metformin therapy
* BMI less than or equal to 39

Exclusion Criteria:

* Type 1 diabetes, diabetes resulting from pancreatic injury or secondary forms of diabetes
* Treatment with thiazolidinediones or use of insulin within the previous 3 months
* Significant illness within 2 weeks prior to dosing
* High fasting triglycerides as defined by the protocol

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-02; Primary Completion 2005-11 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Effect on insulin sensitivity at 6 weeks

SECONDARY OUTCOMES:
Lipolysis rate after 6 weeks of treatment
Plasma free fatty acid concentration after 6 weeks of treatment
Hepatic glucose production after 6 weeks of treatment
Glucose disposal after 6 weeks of treatment
Gluconeogenesis rate after 6 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: David Kelley, MD, Principal Investigator — University of Pittsburgh